CLINICAL TRIAL: NCT00881894
Title: Single-site, Open-label, Randomized, Cross-over Trial to Evaluate the Bioequivalence of Single Dose Rotigotine Transdermal Patch (4.5mg/10cm^2) From 2 Different Manufacturing Processes
Brief Title: Study in Healthy Volunteers to Prove That 2 Rotigotine Patches From Different Manufacturing Processes Deliver Equivalent Drug Amount to the Body.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SP0951
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Results first posted 2009-12-25 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Rotigotine; Neupro®; Transdermal Patch
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A-B (Test: PR2.1.1 - Reference: PR1.0) (Experimental): Two single applications of rotigotine patches from two different manufacturing processes in the order A-B separated by a washout phase of at least 5 days
  Interventions: Drug: Rotigotine transdermal patch
- Sequence B-A (Reference: PR1.0 - Test: PR2.1.1) (Experimental): Two single applications of rotigotine patches from two different manufacturing processes in the order B-A separated by a washout phase of at least 5 days
  Interventions: Drug: Rotigotine transdermal patch

INTERVENTIONS:
Drug: Rotigotine transdermal patch — Rotigotine 4.5mg/10cm^2 patch applied for 24 hours
  Other Names: Neupro®

SUMMARY:
The major aim of this study is to investigate and compare the drug amount delivered to the body after sequential application of 2 rotigotine transdermal patches from 2 different manufacturing processes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy White, male volunteers between 18 and 55 years of age (inclusive).
* BMI between 19 and 28 kg/m² (inclusive).

Exclusion Criteria:

* Previous participation in a clinical study with rotigotine
* History or current condition of epilepsy and/or seizures.
* Known clinically relevant allergy or known/suspected clinically relevant drug hypersensitivity.
* History of significant skin hypersensitivity to adhesives or other transdermal products or recently unresolved contact dermatitis.
* History or present condition of an atopic or eczematous dermatitis, psoriasis, and/or an active skin disease.
* Clinically relevant abnormality in physical examination, ECG, vital signs or safety laboratory examinations.
* Positive HIV, hepatitis B or C test or positive alcohol or drug test.
* Relevant hepatic or renal dysfunction
* Intake of medication that might interfere with the test drug within 2 weeks prior to dosing.
* Thickly hair-covered abdomen resulting in difficulties in finding appropriate patch application sites

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Neuss, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Elshoff JP, Timmermann L, Schmid M, Arth C, Komenda M, Brunnert M, Bauer L. Comparison of the bioavailability and adhesiveness of different rotigotine transdermal patch formulations. Curr Med Res Opin. 2013 Dec;29(12):1657-62. doi: 10.1185/03007995.2013.841666. Epub 2013 Sep 23. PMID 24006953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 52, healthy, male subjects has been randomized in order to complete the trial with at least 44 subjects eligible for the Pharmacokinetic Set (PKS). Baseline characteristics refer to the PKS.
Pre-assignment Details: Patients with an insufficient patch adhesiveness were excluded from the PKS.
Period: Overall Study
Arm/Group | Sequence A-B (Test: PR2.1.1 - Reference: PR1.0) | Sequence B-A (Reference: PR1.0 - Test: PR2.1.1)
Started | 26 | 26
Pharmacokinetic Set (PKS) | 23 (Patients with an insufficient patch adhesiveness were excluded from the PKS.) | 21 (Patients with an insufficient patch adhesiveness were excluded from the PKS.)
Completed | 25 | 23
Not Completed | 1 | 3
Not completed — Consent withdrawn | 0 | 1
Not completed — Other reasons for premature termination | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A-B (Test: PR2.1.1 - Reference: PR1.0) | Sequence B-A (Reference: PR1.0 - Test: PR2.1.1) | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (9.8) | 39.3 (9.1) | 39.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 23 | 21 | 44
Region of Enrollment [Number; unit: participants]
  Germany | 23 | 21 | 44
Weight [Mean (Standard Deviation); unit: kg] | 78.98 (7.08) | 79.98 (8.20) | 79.45 (7.57)

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-tz) of Unconjugated Rotigotine
Description: The AUC(0-tz) is the area under the plasma concentration- time curve from zero up to the last analytically quantifiable concentration.
Time Frame: Pharmacokinetic samples were taken predose, after 1, 2, 3, 4, 6, 8, 12, 16, 24 (before patch removal), 25, 26, 28, 30, 32, 36, 40 and 48 hours after patch application
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*h
Groups:
- Treatment A (Test: PR2.1.1): Rotigotine transdermal patch (4.5 mg/ 10 cm^2) from modified manufacturing process (Test; drug product PR2.1.1); single application of 1 patch for 24 hours
- Treatment B (Reference: PR1.0): Rotigotine transdermal patch (4.5 mg/ 10 cm^2) from originally approved manufacturing process (Reference; drug product PR1.0); single application of 1 patch for 24 hours
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
(ng/ mL)*h | 3.0168 (1.4077) | 3.0635 (1.4309)
Statistical Analysis 1: Comparison: Treatment A (Test: PR2.1.1) vs Treatment B (Reference: PR1.0); Bioequivalence testing by using the 90% Confidence Interval (CI); Test type: Non-Inferiority or Equivalence — If the 90% Confidence Interval for the ratio of geometric LS- Means is included within 0.8- 1.25, the patches are considered bioequivalent; ANOVA; ANOVA for log- transformed values has been used as the basis for calculation of point estimates (LS- Means) and Confidence Intervals (CIs); ratio of geometric LS- Means = 0.9864, 90% CI [0.9103 to 1.0688] — Bioequivalence is concluded if the 90% CIs for the ratio Treatment A/ Treatment B are fully included in the acceptance range from 0.8- 1.25 for AUC(0-tz) and Cmax

2. Primary Outcome: Cmax of Unconjugated Rotigotine
Description: The Cmax is the maximum plasma concentration.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng/ mL
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
ng/ mL | 0.14418 (0.06211) | 0.15155 (0.06540)
Statistical Analysis 1: Comparison: Treatment A (Test: PR2.1.1) vs Treatment B (Reference: PR1.0); Bioequivalence testing by using the 90% Confidence Interval (CI); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of geometric LS- Means = 0.9584, 90% CI [0.8861 to 1.0367] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUC(0-∞) of Unconjugated Rotigotine
Description: The AUC(0-∞) is the area under the plasma concentration- time curve from zero up to infinity.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*h
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
(ng/ mL)*h | 3.12622 (1.41536) | 3.16403 (1.43028)
Statistical Analysis 1: Comparison: Treatment A (Test: PR2.1.1) vs Treatment B (Reference: PR1.0); Bioequivalence testing by using the 90% Confidence Interval (CI); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of geometric LS- Means = 0.9896, 90% CI [0.9179 to 1.0671]

4. Secondary Outcome: AUC(0-tz)Norm (Apparent Dose) of Unconjugated Rotigotine
Description: The AUC(0-tz)Norm (Apparent dose) is the area under the plasma concentration- time curve from zero up to the last analytically quantifiable concentration normalized by apparent dose (mg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*(h/ mg)
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
(ng/ mL)*(h/ mg) | 1.78200 (0.71912) | 1.58900 (0.54806)

5. Secondary Outcome: AUC(0-tz)Norm (BW) of Unconjugated Rotigotine
Description: The AUC(0-tz)Norm (BW) is the area under the plasma concentration- time curve from zero up to the last analytically quantifiable concentration normalized by body weight (kg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*h*kg
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
(ng/ mL)*h*kg | 239.241 (112.475) | 243.841 (116.640)

6. Secondary Outcome: Cmax,Norm (Apparent Dose) of Unconjugated Rotigotine
Description: The Cmax,Norm (Apparent dose) is the maximum plasma concentration normalized by apparent dose.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL) / mg
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
(ng/ mL) / mg | 0.085822 (0.032789) | 0.079619 (0.027178)

7. Secondary Outcome: Cmax,Norm (BW) of Unconjugated Rotigotine
Description: The Cmax,Norm (BW) is the maximum plasma concentration normalized by body weight (kg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*kg
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
(ng/ mL)*kg | 11.4391 (4.9667) | 12.0441 (5.3133)

8. Secondary Outcome: Tmax of Unconjugated Rotigotine
Description: The Tmax is the time to reach a maximum plasma concentration after patch application.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
hour (h) | 16.00 (6.18) [8.0 to 28.0] | 16.00 (5.26) [6.0 to 26.0]

9. Secondary Outcome: MRT of Unconjugated Rotigotine
Description: The MRT is the mean residence time.
Time Frame: Pharmacokinetic samples were taken predose, after 1, 2, 3, 4, 6, 8, 12, 16, 24(before patch removal), 25, 26, 28, 30, 32, 36, 40 and 48 hours after patch application.
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
hour (h) | 19.012 (1.809) | 18.882 (1.802)

10. Secondary Outcome: λz of Unconjugated Rotigotine
Description: The λz is the rate constant of elimination.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: 1/ hour (1/h)
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
1/ hour (1/h) | 0.153848 (0.037525) | 0.151239 (0.025301)

11. Secondary Outcome: t1/2 of Unconjugated Rotigotine
Description: The t1/2 is the terminal half- life.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
hour (h) | 4.7665 (1.1499) | 4.7128 (0.8088)

12. Secondary Outcome: CL/f of Unconjugated Rotigotine
Description: The CL/f is the apparent total body clearance.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: L/ h
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
L/ h | 1825.38 (1058.21) | 1822.13 (1060.42)

13. Secondary Outcome: Apparent Dose
Description: Apparent dose of unconjugated rotigotine in mg. The Apparent dose of unconjugated rotigotine was determined from the patches removed on Day 2.
Time Frame: 48 hours
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Number analyzed (Participants) | 44 | 44
mg | 1.676 (0.423) | 1.890 (0.561)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected within 48 hours.
Description: Adverse events are reported for the Safety Set (SS). The SS includes all randomized subjects who received at least 1 dose of trial medication (N=52). Two subjects terminated the study prematurely after period 1 (1 subject in sequence A-B and 1 in sequence B-A). Therefore the number of subject exposed to each treatment is N=51.
Arm/Group | Treatment A (Test: PR2.1.1) | Treatment B (Reference: PR1.0)
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 21/51 | 21/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (Test: PR2.1.1) (N=51) | Treatment B (Reference: PR1.0) (N=51)
Abnormal Sensation in Eye (Eye disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Application Site Pruritus (General disorders) | 12 (12) | 12 (12)
Application Site Cold Feeling (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (9) | 5 (5)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3)
Syncope Vasovagal (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Disturbance in Attention (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.